CLINICAL TRIAL: NCT01005901
Title: A 26-week Treatment, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of NVA237 in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of NVA237 Versus Placebo
Acronym: GLOW 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237A2304; 2009-013504-32 (EudraCT Number)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; NVA; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Glycopyrronium bromide (Experimental): Glycopyrronium bromide 50µg delivered once daily via Single Dose Dry Powder Inhaler (SDDPI). At visit 1 all patients were provided with a short acting β2-agonist (salbutamol/albuterol) which they were instructed to use throughout the study as rescue medication.
  Interventions: Drug: Glycopyrronium bromide
- Placebo (Placebo Comparator): Placebo delivered once daily via SDDPI. At Visit 1 all patients were provided with a short acting β2-agonist (salbutamol/albuterol) which they were instructed to use throughout the study as rescue medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glycopyrronium bromide — Glycopyrronium bromide 50µg was supplied as inhalation capsules for use via a Single Dose Dry Powder Inhaler (SDDPI)
  Arms: Glycopyrronium bromide
Drug: Placebo — Placebo inhalation capsules were provided for use via a SDDPI
  Arms: Placebo

SUMMARY:
A study to assess the safety, tolerability and efficacy of NVA237 versus placebo in patients with moderate-to-severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2008) and:

* Smoking history of at least 10 pack-years
* Post-bronchodilator FEV1 < 80% and ≥ 30% of the predicted normal value
* Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion Criteria:

1. Patients who have had a lower respiratory tract infection within 6 weeks prior to Visit 1
2. Patients with concomitant pulmonary disease
3. Patients with a history of asthma
4. Any patient with lung cancer or a history of lung cancer
5. Patients with a history of certain cardiovascular comorbid conditions
6. Patients with a known history and diagnosis of alpha-1 antitrypsin deficiency
7. Patients in the active phase of a supervised pulmonary rehabilitation program
8. Patients contraindicated for tiotropium or ipratropium treatment or who have shown an untoward reaction to inhaled anticholinergic agents Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1324 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (96):
- United States (33):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fairhope, Alabama
  - Novartis Investigative Site, Glendale, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Madisonville, Kentucky
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Biddeford, Maine
  - Novartis Investigative Site, Pikesville, Maryland
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Bellevue, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Lincoln, Rhode Island
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Corpus Christi, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Richmond, Virginia
- Novartis Investigative Site, Daw Park SA, Australia
- Canada (7):
  - Novartis Investigative Site, Bridgewater, Nova Scotia
  - Novartis Investigative Site, Courtice, Ontario
  - Novartis Investigative Site, Mississuaga, Ontario
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Japan (19):
  - Novartis Investigative Site, Asahikawa
  - Novartis Investigative Site, Hamakita
  - Novartis Investigative Site, Himeji
  - Novartis Investigative Site, Hitachi
  - Novartis Investigative Site, Kishiwada
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Matsue
  - Novartis Investigative Site, Matsusaka
  - Novartis Investigative Site, Moriya
  - Novartis Investigative Site, Naka-gun
  - Novartis Investigative Site, Obihiro
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Ōta-ku
  - Novartis Investigative Site, Ōtsu
  - Novartis Investigative Site, Sapporo
  - Novartis Investigative Site, Takatsuki
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Yabu
  - Novartis Investigative Site, Yonezawa
- Netherlands (5):
  - Novartis Investigative Site, Almelo
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Harderwijk
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Zutphen
- Romania (3):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Iași
  - Novartis Investigative Site, Timișoara
- Russia (9):
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Sochy
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Pusan
  - Novartis Investigative site, Seoul
- Spain (6):
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Canet de Mar
  - Novartis Investigative Site, Cáceres
  - Novartis Investigative Site, Centelles
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (9):
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Diyarbakır
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kinikli/Denizli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Soke/Aydin
  - Novartis Investigative Site, Yenisehir/Izmir

REFERENCES:
- [Result] D'Urzo A, Ferguson GT, van Noord JA, Hirata K, Martin C, Horton R, Lu Y, Banerji D, Overend T. Efficacy and safety of once-daily NVA237 in patients with moderate-to-severe COPD: the GLOW1 trial. Respir Res. 2011 Dec 7;12(1):156. doi: 10.1186/1465-9921-12-156. PMID 22151296
- [Derived] D'Urzo A, Kerwin E, Overend T, D'Andrea P, Chen H, Goyal P. Once daily glycopyrronium for the treatment of COPD: pooled analysis of the GLOW1 and GLOW2 studies. Curr Med Res Opin. 2014 Mar;30(3):493-508. doi: 10.1185/03007995.2013.858618. Epub 2013 Nov 19. PMID 24156566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1324 participants were screened. 822 participants entered the study.
Period: Overall Study
Arm/Group | Glycopyrronium Bromide | Placebo
Started | 552 | 270
Safety Population | 550 | 267
Full Analysis Set | 534 | 260
Completed | 450 | 212
Not Completed | 102 | 58
Not completed — Withdrawal by Subject | 38 | 14
Not completed — Adverse Event | 30 | 16
Not completed — Administrative problems | 21 | 13
Not completed — Unsatisfactory therapeutic effect | 5 | 5
Not completed — Protocol Violation | 4 | 3
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Patient's inability to use the device | 1 | 1
Not completed — No longer requires study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycopyrronium Bromide | Placebo | Total
Number analyzed (Participants) | 550 | 267 | 817
Age, Customized [Number; unit: participants] — All baseline measures are based on safety population.
  participants
    <65 years | 278 | 134 | 412
    65 to <75 years | 199 | 98 | 297
    >=75 years | 73 | 35 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 52 | 148
  Male | 454 | 215 | 669

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at 12 Weeks
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 hour 15 minute and 23 hour 45 minute post-dose FEV1 readings. Mixed model used baseline FEV1,baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) The FAS included all randomized patients who received at least one dose of study medication. Patients in this group were analyzed according to the treatment to which they were randomized. Missing trough FEV1 values at week 12 were imputed using LOCF with pre-dose trough FEV1.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 512 | 243
Liters | 1.408 (0.0105) | 1.301 (0.0137)

2. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score After 26 Weeks of Treatment
Description: Transition Dyspnea Index (TDI) captures changes from baseline. The TDI score is based on three domains with each domain scored from -3 (major deterioration) to +3 (major improvement), to give an overall score of -9 to +9, a negative score indicating a deterioration from baseline. A TDI focal score of 1 is considered to be a clinically significant improvement from baseline. Mixed model used baseline TDI, baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: 26 weeks
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication. Patients per treatment group with no missing data were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 493 | 240
Units on a scale | 1.84 (0.257) | 0.80 (0.294)

3. Secondary Outcome: Quality of Life Assessment With St. George's Respiratory Questionnaire (SGRQ) Total Score After 26 Weeks of Treatment
Description: SGRQ is a health related quality of life questionnaire consisting of 51 items in three components: symptoms, activity, and impacts. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life. Mixed model used baseline SGRQ, baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: 26 weeks
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication. Individual component score was imputed with LOCF (last observation carried forward).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 502 | 246
Units on a scale | 39.50 (0.813) | 42.31 (0.992)

4. Secondary Outcome: Time to First Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation During 26 Weeks of Treatment
Description: The time to the first moderate or severe COPD exacerbation was the study day on which the patient experienced first moderate or severe COPD exacerbation. COPD exacerbations are considered to be moderate if treatment with systemic corticosteroids and/or antibiotics was required. COPD exacerbations are considered to be severe if treatment for moderate severity and hospitalization were required.
Time Frame: 26 weeks
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication.
  The median values were not estimable.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 534 | 260
Days | NA [NA to NA] — The median values were not estimable because less than 50% of patients had a moderate or severe COPD exacerbation during the study. | NA [NA to NA] — The median values were not estimable because less than 50% of patients had a moderate or severe COPD exacerbation during the study.

5. Secondary Outcome: Change From Baseline in the Mean Number of Puffs Per Day of Rescue Medication Over the Study Duration (Baseline to Week 26)
Description: Participants recorded the number of puffs of rescue medication taken in the previous 12 hours in the morning and evening. The total number of puffs of rescue medication per day over the full 26 weeks was calculated and divided by the total number of days with non-missing rescue medication data to derive the mean daily number of puffs of rescue medication taken for the patient.
Time Frame: 26 weeks
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication. Patients with observations both at baseline and week 26 were included in this analysis
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 529 | 259
Puffs per day | -1.21 (0.122) | -0.75 (0.156)

6. Secondary Outcome: FEV1 at Each Time-point on Day 1 and Week 26
Description: Spirometry was conducted according to internationally accepted standards. FEV1 was measured at all time points up to 4 hours post-dose, and at 23 hours 15 min and 23 hours 45 min, by visit. Mixed model used baseline FEV1,baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: Day 1 and Week 26
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication. "n" indicates number of patients with observation at each time-point
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 519 | 253
Liters
  Day 1: 5 min (n = 497, 240) | 1.388 (0.0057) | 1.295 (0.0076)
  Day 1: 15 min (n = 503, 249) | 1.435 (0.0066) | 1.292 (0.0087)
  Day 1: 30 min (n = 511, 252) | 1.472 (0.0070) | 1.299 (0.0093)
  Day 1: 1 hour (n = 513, 253) | 1.493 (0.0070) | 1.296 (0.0094)
  Day 1: 2 hours (n = 514, 251) | 1.562 (0.0076) | 1.355 (0.0102)
  Day 1: 3 hours (n = 519, 248) | 1.544 (0.0079) | 1.349 (0.0108)
  Day 1: 4 hours (n = 514, 247) | 1.548 (0.0077) | 1.365 (0.0105)
  Day 1: 23 hours 15 min (n = 499, 244) | 1.400 (0.0078) | 1.289 (0.0103)
  Day 1: 23 hours 45 min (n = 498, 244) | 1.428 (0.0083) | 1.328 (0.0108)
  Week 26: pre-dose trough (n = 447, 208) | 1.371 (0.0100) | 1.256 (0.0140)
  Week 26: -45 min (n = 447, 208) | 1.373 (0.0104) | 1.256 (0.0145)
  Week 26: -15 min (n = 443, 205) | 1.368 (0.0104) | 1.252 (0.0144)
  Week 26: 5 min (n = 439, 208) | 1.409 (0.0106) | 1.255 (0.0147)
  Week 26: 15 min (n = 435, 205) | 1.427 (0.0109) | 1.269 (0.0152)
  Week 26: 30 min (n = 440, 207) | 1.433 (0.0112) | 1.259 (0.0155)
  Week 26: 1 hour (n = 438, 206) | 1.459 (0.0115) | 1.251 (0.0159)
  Week 26: 2 hours (n = 438, 203) | 1.508 (0.0114) | 1.299 (0.0160)
  Week 26: 3 hours (n = 439, 204) | 1.504 (0.0124) | 1.299 (0.0170)
  Week 26: 4 hours (n = 438, 205) | 1.489 (0.0114) | 1.312 (0.0158)
  Week 26: 23 hours 15 min (n = 434, 206) | 1.386 (0.0118) | 1.267 (0.0158)
  Week 26: 23 hours 45 min (n = 434, 206) | 1.396 (0.0116) | 1.282 (0.0157)

7. Secondary Outcome: Forced Vital Capacity (FVC) at Each Time-point on Day 1 and Week 26
Description: Spirometry was conducted according to internationally accepted standards. FVC was calculated at each time point up to 4 hours post-dose and at 23 hours 15 min and 23 hours 45 min, by visit. Mixed model used baseline FVC, baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: Day 1 and Week 26
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 534 | 260
Liters
  Day 1: 5 min (n = 497, 240) | 2.887 (0.0132) | 2.675 (0.0173)
  Day 1: 15 min (n = 503, 249) | 2.943 (0.0147) | 2.660 (0.0188)
  Day 1: 30 min (n = 511, 252) | 2.948 (0.0155) | 2.637 (0.0199)
  Day 1: 1hour (n = 513, 253) | 3.019 (0.0148) | 2.669 (0.0198)
  Day 1: 2 hours (n = 514, 251) | 3.086 (0.0166) | 2.754 (0.0219)
  Day 1: 3 hours (n = 519, 248) | 3.096 (0.0168) | 2.783 (0.0227)
  Day 1: 4 hours (n = 514, 247) | 3.064 (0.0161) | 2.760 (0.0217)
  Day 1: 23 hours 15 min (n = 499, 244) | 2.895 (0.0169) | 2.693 (0.0221)
  Day 1: 23 hours 45 min (n = 498, 244) | 2.907 (0.0169) | 2.718 (0.0219)
  Week 26: Pre-dose trough (n = 447, 208) | 2.827 (0.0238) | 2.623 (0.0305)
  Week 26: -45 min (n = 447, 208) | 2.859 (0.0271) | 2.658 (0.0337)
  Week 26: -15 min (n = 443, 205) | 2.798 (0.0235) | 2.589 (0.0306)
  Week 26: 5 min (n = 439, 208) | 2.891 (0.0251) | 2.639 (0.0318)
  Week 26: 15 min (n = 435, 205) | 2.895 (0.0240) | 2.660 (0.0309)
  Week 26: 30 min (n = 440, 207) | 2.885 (0.0239) | 2.603 (0.0310)
  Week 26: 1 hour (n = 438, 206) | 2.938 (0.0256) | 2.625 (0.0329)
  Week 26: 2 hours (n = 438, 203) | 2.977 (0.0225) | 2.687 (0.0302)
  Week 26: 3 hours (n = 439, 204) | 3.016 (0.0270) | 2.742 (0.0345)
  Week 26: 4 hours (n = 438, 205) | 2.962 (0.0225) | 2.709 (0.0303)
  Week 26: 23 hours 15 min (n = 434, 206) | 2.884 (0.0257) | 2.673 (0.0322)
  Week 26: 23 hours 45 min (n = 434, 206) | 2.859 (0.0234) | 2.669 (0.0306)

8. Secondary Outcome: FEV1 Area Under the Curve (AUC) (5 Min - 12 Hour) at Day 1, Week 12 and Week 26
Description: The standardized (with respect to the length of time) area under the curve (AUC) for FEV1 was calculated using trapezoidal rule between 5 min and 12 h post dose at Week 1 Day 1, Week 12 and Week 26 for every patient in the serial spirometry subgroup. Mixed model used baseline FEV1,baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: Day 1, Week 12 and Week 26
Population: Serial spirometry group, a sub-set of the full analysis set of patients. Twelve hour serial spirometry was conducted in this subset of patients in selected centers at Day 1. At week 12/13 and week 26/27 a 24 hour serial spirometry was performed. "n" is the number of patients with non-missing observations at each time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 169 | 83
Liters
  Day 1 (n = 169, 83) | 1.475 (0.0129) | 1.320 (0.0173)
  Week 12 (n = 153, 75) | 1.433 (0.0179) | 1.284 (0.0244)
  Week 26 (n = 149, 70) | 1.445 (0.0199) | 1.238 (0.0274)

9. Secondary Outcome: FEV1 Area Under Curve (AUC) (5 Min - 23 Hour 45 Min) at Week 12 and Week 26
Description: The standardized (with respect to the length of time) area under the curve (AUC) for FEV1 was calculated using trapezoidal rule between 5 min and 23 h 45 min post dose at week12/week 13and week 26/week 27 where available for every patient in the serial spirometry subgroup. Mixed model used baseline FEV1,baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: Week 12 and Week 26
Population: Serial spirometry group, a sub-set of the full analysis set of patients. Twelve hour serial spirometry was conducted in this subset of patients in selected centers at Day 1. At week 12/13 and week 26/27 a 24 hour serial spirometry was performed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 169 | 83
Liters
  Week 12 (n = 153, 75) | 1.401 (0.0167) | 1.268 (0.0228)
  Week 26 (n = 149, 70) | 1.412 (0.0185) | 1.213 (0.0254)

10. Secondary Outcome: Trough FEV1 and FVC at Day 1 and Week 26
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 hour 15 minute and 23 hour 45 minute post-dose FEV1 readings. Mixed model used baseline FEV1, baseline ICS use, FEV1 prior to inhalation of SABA, and FEV1 45 minutes post-inhalation of SABA as covariates.
  Trough FVC was defined as the average of the 23 hour 15 minute and 23 hour 45 minute post-dose FVC readings. Mixed model used baseline FVC, baseline ICS use, FEV1 prior to inhalation of SABA, and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: Day 1 and Week 26
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication. If one of the 23 h 15 min or 23 h 45 min values are missing then the remaining non-missing value is taken as trough FEV1 or trough FVC. If both values are missing, then their trough FEV1 or trough FVC is regarded as missing
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 534 | 260
Liters
  Day 1: FEV1 (n = 508, 248) | 1.414 (0.0075) | 1.309 (0.0099)
  Week 26: FEV1 (n = 461, 217) | 1.387 (0.0112) | 1.275 (0.0150)
  Day 1: FVC (n = 508, 248) | 2.901 (0.0154) | 2.705 (0.0202)
  Week 26: FVC (n = 438, 208) | 2.867 (0.0236) | 2.668 (0.0300)

11. Secondary Outcome: Change in 24-hourly Mean Heart Rate at Day 1, Week 12 and Week 26
Description: The mean heart rate was collected with a 24 hour Holter monitor in a sub-set of the safety population. The change between baseline and day 1, week 12 and week 26 was calculated. The analysis of the Holter recordings was performed by a central facility. Data on heart rate, heart rate variability, supraventricular and ventricular ectopy were collected and assessed.
Time Frame: Baseline, Day 1, Week 12 and Week 26
Population: The safety set included all patients who received at least one dose of study medication whether or not being randomized. A sub-set of the safety population had 24 hour Holter monitoring. "n" indicates patients with observations both at baseline and each endpoint.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 42 | 23
beats per minute
  Day 1: (n = 42, 23) | -1.77 (7.583) | -1.28 (8.676)
  Week 12: (n = 42, 20) | -1.99 (7.489) | -1.70 (7.230)
  Week 26: (n = 37, 22) | -4.40 (9.347) | -2.60 (9.349)

12. Secondary Outcome: Number of Participants With Adverse Events, Death, and Serious or Clinically Significant Adverse Events or Related Discontinuations
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: 26 Weeks and 30 Day follow-up
Population: The safety set included all patients who received at least one dose of study medication whether or not being randomized. Patients were randomized according to the treatment they received.
Measure: Number; unit: participants
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 550 | 267
participants
  Participants with at least one AE | 317 | 174
  Death | 3 | 3
  SAE(s) | 41 | 24
  Discontinuation due to AE(s) | 32 | 19
  Discontinuation due to SAE(s) | 15 | 8
  Discontinuation due to non-SAE(s) | 18 | 11
  AE leading to dose interruption | 12 | 8
  AE requiring significant additional therapy | 246 | 155
  AE leading to new or prolonged hospitalization | 35 | 21

13. Secondary Outcome: Rate of Moderate or Severe COPD Exacerbations Over the 26 Week Treatment Period
Description: One overall rate is calculated for the entire study population. Rate is the number of moderate or severe exacerbations per year = total number of moderate or severe exacerbations for all participants/total number of treatment years for all participants. COPD exacerbations were considered to be moderate if treatment with systemic corticosteroids and/or antibiotics was required. COPD exacerbations were considered to be severe if treatment for moderate severity and hospitalization were required.
Time Frame: 26 weeks
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication.
Measure: Number; unit: exacerbations per year
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 534 | 260
exacerbations per year | 0.43 | 0.59

14. Secondary Outcome: Percentage of Nights With no Nighttime Awakenings Over the 26 Week Treatment Period
Description: The percentage of nights with no nighttime awakenings is defined as the total number of nights with no nighttime awakenings over the 26 week treatment period divided by the total number of night where diary recordings have been made.
  Mixed model used baseline nighttime awakenings, baseline ICS use, FEV1 prior to inhalation of SABA, and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: 26 Weeks
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication. At 26 weeks, the analysis is based on only patients with a value at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of nights with no awakenings
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 527 | 258
percentage of nights with no awakenings | 55.96 (1.537) | 54.37 (1.970)

15. Secondary Outcome: Percentage of Days With no Daytime Symptoms Over the 26 Week Treatment Period
Description: The percentage of days with no daytime symptoms is defined as the total number of days with no daytime symptoms over the 26 week treatment period divided by the total number of days where diary recordings have been made.
  Mixed model used baseline daytime symptoms, baseline ICS use, FEV1 prior to inhalation of SABA, and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: 26 Weeks
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: percentage of days with no symptoms
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 528 | 258
percentage of days with no symptoms | 5.70 (0.799) | 5.78 (1.076)

16. Secondary Outcome: Percentage of Days Able to Perform Usual Daily Activities Over the 26 Week Treatment Period
Description: The percentage of days able to perform usual daily activities is defined as the total number of days able to perform usual activities over the 26 week treatment period divided by the total number of days where diary recordings have been made.
  Mixed model used baseline ability to perform usual daily activities, baseline ICS use, FEV1 prior to inhalation of SABA, and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: 26 Weeks
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 528 | 258
percentage of days | 40.31 (1.473) | 35.19 (1.907)

17. Secondary Outcome: Mean Daily Total Symptom Score Over the 26 Week Treatment Period
Description: The daily symptom score was calculated as the sum of the worst of the morning and evening assessments for each symptom (symptoms, cough, wheeze, sputum color/production, and breathlessness). The score can range from 0 to 18 with 0 indicating no symptoms. The higher the score, the worse the symptomatic status. A negative change (lower number) indicates improvement.
  Mixed model used baseline symptom variables, baseline inhaled corticosteroid (ICS) use, FEV1 prior to inhalation of short acting beta-agonist (SABA), and FEV1 45 minutes post-inhalation of SABA as covariates.
Time Frame: 26 Weeks
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Glycopyrronium Bromide | Placebo
Number analyzed (Participants) | 534 | 260
units on a scale | -1.54 (0.097) | -1.18 (0.129)

ADVERSE EVENTS:
Arm/Group | Glycopyrronium Bromide | Placebo
Serious Adverse Events (participants affected / at risk) | 41/550 | 24/267
Other Adverse Events (participants affected / at risk) | 132/550 | 85/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrronium Bromide (N=550) | Placebo (N=267)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Cataract (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 3 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrronium Bromide (N=550) | Placebo (N=267)
Nasopharyngitis (Infections and infestations) | 28 | 21
Upper respiratory tract infection (Infections and infestations) | 23 | 20
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 105 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.